CLINICAL TRIAL: NCT06754787
Title: Renal Recovery After PEEP Weaning in ARDS
Brief Title: Renal Recovery After PEEP Weaning in ARDS (RE2SDRA)
Acronym: RE2SDRA
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0031 - RE2SDRA
Record Dates: First submitted 2024-12-11; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-10

CONDITIONS: ARDS (Acute Respiratory Distress Syndrome); AKI - Acute Kidney Injury
MeSH Terms: conditions — Acute Lung Injury; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to investigate renal recovery in ARDS after PEEP weaning. The primary outcome was the variation of the hourly urine output (HUO), 48 h after PEEP weaning. Secondary outcomes were the need for RRT and mortality. Two groups were defined depending wether hourly urine output was greater or lower than 0.35 mL/kg/h.

ELIGIBILITY:
Inclusion Criteria:

* intubated for more than 48 hours, exposed to a PEEP≥ 8 cmH20

Exclusion Criteria:

* chronic end-stage renal disease on admission
* refusal to participate
* non-opposition could not be obtained from themselves or their trusted support person in the event of incapacity
* under legal protection.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients were included if they were intubated for more than 48 hours, exposed to a PEEP≥ 8 cmH20 followed by a successful PEEP weaning defined as ≤6 cmH20 for more than 72 hours.
  Patients were excluded if they had chronic end-stage renal disease on admission, refusal to participate, whose non-opposition could not be obtained from themselves or their trusted support person in the event of incapacity or if they were under legal protection.
  Patients with impaired hourly urine output (HUO) (≤ 1 ml/kg/h) before PEEP weaning were selected.
  Therefore, 120 patients of a cohort of 338 who required invasive mechanical ventilation for ARDS in the ICU of the Brest University Hospital were included.
  The ethics committee of Brest university hospital approved the investigation RE2SDRA on 03/14/2024.
  No additional diagnostic, treatment or monitoring procedures were conducted.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2024-03-21 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Variation of the hourly urine output on day 2 after PEEP weaning | From enrollement to day 2 after PEEP weaning
  Variation of the hourly urine output on day 2 after PEEP weaning

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement

REFERENCES:
- See also: Related Info — https://doi.org/10.3389/fped.2021.744110
- See also: Related Info — https://doi.org/10.1097/CCM.0000000000003832
- See also: Related Info — https://doi.org/10.1186/s12882-019-1439-2